CLINICAL TRIAL: NCT02373306
Title: Non-invasive Programmed Stimulation to Identify High-risk Patients With Implanted Cardioverter-defibrillator
Brief Title: NIPS to Identify High-risk Patients With ICD
Acronym: NIPS-ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Centre, Poland (Other)
Responsible Party: Principal Investigator, Piotr Futyma, MD, St. Joseph's Centre, Poland
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NIPS-ICD
Record Dates: First submitted 2014-12-23; First posted 2015-02-27 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Malignant Arrhythmia
Keywords: Risk stratification; ICD intervention; occurrence during one-year follow-up after NIPS
MeSH Terms: interventions — Sulfamethazine

ARMS (2):
- NIPS-sensitive group (Active Comparator): Patients who had sustained or hemodynamically unstable arrhythmia induction during non-invasive programmed stimulation.
  Interventions: Procedure: Sustained or hemodynamically unstable arrhythmia induction during non-invasive programmed stimulation
- Control group (No Intervention): Patients who had no sustained or hemodynamically unstable arrhythmias induction during non-invasive programmed stimulation.

INTERVENTIONS:
Procedure: Sustained or hemodynamically unstable arrhythmia induction during non-invasive programmed stimulation
  Arms: NIPS-sensitive group

SUMMARY:
Implantable cardioverter-defibrillator (ICD) is a widely used and effective therapy which reduces the risk of cardiac death in many cardiac diseases, both implanted for secondary and primary prevention. It is known that recurrent arrhythmias and ICD discharges have adverse prognostic significance. Parameters that would identify patients who are at increased risk of arrhythmias and appropriate ICD interventions would be of clinical value. The aim of the study is to evaluate the usefulness of non-invasive programmed stimulation (NIPS) in determining the likelihood of life-threatening arrhythmic events in patients with ICD.

DETAILED DESCRIPTION:
Some studies have shown that factors predicting ventricular tachycardia (VT) or ventricular fibrillation (VF) recurrences and consequently ICD interventions, include patient's age, New York Heart Association class heart failure, left ventricular ejection fraction (LVEF), the presence of atrial fibrillation (AF), the QRS complex width, and the status of renal function. However, the accuracy of these parameters is limited and other variables that may identify vulnerable patients are sought. This may have important clinical implications because such patients could receive more aggressive antiarrhythmic therapy or may undergo prophylactic ablation of arrhythmia substrate to prevent the occurrence of arrhythmias and ICD discharges. Indeed, some studies suggested that it might be worth to perform prophylactic ablation of VT in patients with previously implanted ICD, however, this approach has not entered into daily clinical practice.

One of the methods of risk stratification for sudden cardiac death which has been used for many years, is programmed ventricular stimulation (PVS). This is an invasive study assessing the likelihood of VT or VF induced by stimulation to occur. This test has been also used in order to qualify for prophylactic ICD implantation in patients with LVEF 31-40% and non-sustained VT in ambulatory ECG. The primary disadvantage of PVS is its invasiveness. Modern ICDs are relatively complex devices with a number of functions, including the possibility to perform NIPS with implanted electrode located in the right ventricle. NIPS is readily available, inexpensive, minimally burdening ICD battery and less disturbing to the patient, because it does not require any invasive procedure.

Some studies suggested that appropriate interventions occur more frequently in patients who had ventricular arrhythmias induced by NIPS, but prognostic significance of NIPS has not yet been determined. One of the first NIPS-related studies demonstrated that VF/VT inducibility during the test of the device can help to optimize ICD programming, however, predictive value of NIPS had not been studied at that time. In another study, one of the first and few on the prognostic value of NIPS, it has been shown that induction of monomorphic, especially relatively slow VT (cycle length> 280ms) was prognostic for recurrence of arrhythmias. This study was relatively small, the distribution of etiology had not been considered, and some of the results were surprising, eg. previous myocardial infarction of inferior wall, rather than the anterior wall, predicted altered outcome, while LVEF had no prognostic value. In addition, these studies had been carried out many years ago, when the use of primary angioplasty for acute myocardial infarction was low, and therefore the clinical characteristics of the patient groups from that period are different than those of contemporary patients.

ELIGIBILITY:
Inclusion Criteria:

- patients with an ICD implanted both for primary and secondary prevention, regardless of etiology, who are followed in the outpatient clinic of our center, and who do not meet the exclusion criteria

Exclusion Criteria:

* lack of consent for NIPS
* decompensated heart failure
* unstable angina
* persistent/long standing AF without effective anticoagulation (risk of sinus rhythm return during NIPS)
* thrombus in the left ventricle
* appropriate device interventions during the 40 days prior to planned NIPS
* pacing/sensing problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with appropriate intervention of ICD | up to 1 year from date of randomization
  Appropriate intervention of ICD due to ventricular arrhythmia

SECONDARY OUTCOMES:
Number of participants with sudden cardiac (arrhythmic) death | up to 1 year from date of randomization
  Death due to sustained VT/VF, or in the absence of available documentation - death which occurred within one hour of the onset of symptoms

OTHER OUTCOMES:
Number of participants with death from cardiovascular causes | up to 1 year from date of randomization
  Death due to VF, extensive myocardial infarction, electromechanical dissociation, asystole, or end-stage heart failure.
Number of participants with hospitalization for cardiovascular causes | up to 1 year from date of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kułakowski, MD, PhD, FESC, Study Chair — Postgraduate Medical School, Warsaw; Piotr Futyma, MD, Principal Investigator — St. Joseph's Centre, Rzeszów
Locations (1):
- St. Joseph's Centre, Rzeszów, Subcarpathian District, Poland

REFERENCES:
- [Background] Moss AJ, Hall WJ, Cannom DS, Daubert JP, Higgins SL, Klein H, Levine JH, Saksena S, Waldo AL, Wilber D, Brown MW, Heo M. Improved survival with an implanted defibrillator in patients with coronary disease at high risk for ventricular arrhythmia. Multicenter Automatic Defibrillator Implantation Trial Investigators. N Engl J Med. 1996 Dec 26;335(26):1933-40. doi: 10.1056/NEJM199612263352601. PMID 8960472
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Zipes DP, Camm AJ, Borggrefe M, Buxton AE, Chaitman B, Fromer M, Gregoratos G, Klein G, Moss AJ, Myerburg RJ, Priori SG, Quinones MA, Roden DM, Silka MJ, Tracy C, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL, Smith SC Jr, Jacobs AK, Adams CD, Antman EM, Anderson JL, Hunt SA, Halperin JL, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 guidelines for management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: a report of the American College of Cardiology/American Heart Association Task Force and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Develop guidelines for management of patients with ventricular arrhythmias and the prevention of sudden cardiac death) developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Europace. 2006 Sep;8(9):746-837. doi: 10.1093/europace/eul108. Epub 2006 Aug 25. No abstract available. PMID 16935866
- [Background] Tung R, Zimetbaum P, Josephson ME. A critical appraisal of implantable cardioverter-defibrillator therapy for the prevention of sudden cardiac death. J Am Coll Cardiol. 2008 Sep 30;52(14):1111-21. doi: 10.1016/j.jacc.2008.05.058. PMID 18804736
- [Background] Lee DS, Tu JV, Austin PC, Dorian P, Yee R, Chong A, Alter DA, Laupacis A. Effect of cardiac and noncardiac conditions on survival after defibrillator implantation. J Am Coll Cardiol. 2007 Jun 26;49(25):2408-15. doi: 10.1016/j.jacc.2007.02.058. Epub 2007 Jun 11. PMID 17599603
- [Background] Borne RT, Varosy PD, Masoudi FA. Implantable cardioverter-defibrillator shocks: epidemiology, outcomes, and therapeutic approaches. JAMA Intern Med. 2013 May 27;173(10):859-65. doi: 10.1001/jamainternmed.2013.428. PMID 23546173
- [Background] Bigger JT Jr. Prophylactic use of implanted cardiac defibrillators in patients at high risk for ventricular arrhythmias after coronary-artery bypass graft surgery. Coronary Artery Bypass Graft (CABG) Patch Trial Investigators. N Engl J Med. 1997 Nov 27;337(22):1569-75. doi: 10.1056/NEJM199711273372201. PMID 9371853
- [Background] Hohnloser SH, Kuck KH, Dorian P, Roberts RS, Hampton JR, Hatala R, Fain E, Gent M, Connolly SJ; DINAMIT Investigators. Prophylactic use of an implantable cardioverter-defibrillator after acute myocardial infarction. N Engl J Med. 2004 Dec 9;351(24):2481-8. doi: 10.1056/NEJMoa041489. PMID 15590950
- [Background] Buxton AE, Lee KL, Fisher JD, Josephson ME, Prystowsky EN, Hafley G. A randomized study of the prevention of sudden death in patients with coronary artery disease. Multicenter Unsustained Tachycardia Trial Investigators. N Engl J Med. 1999 Dec 16;341(25):1882-90. doi: 10.1056/NEJM199912163412503. PMID 10601507
- [Background] Desai AS, Fang JC, Maisel WH, Baughman KL. Implantable defibrillators for the prevention of mortality in patients with nonischemic cardiomyopathy: a meta-analysis of randomized controlled trials. JAMA. 2004 Dec 15;292(23):2874-9. doi: 10.1001/jama.292.23.2874. PMID 15598919
- [Background] Steinbeck G, Andresen D, Seidl K, Brachmann J, Hoffmann E, Wojciechowski D, Kornacewicz-Jach Z, Sredniawa B, Lupkovics G, Hofgartner F, Lubinski A, Rosenqvist M, Habets A, Wegscheider K, Senges J; IRIS Investigators. Defibrillator implantation early after myocardial infarction. N Engl J Med. 2009 Oct 8;361(15):1427-36. doi: 10.1056/NEJMoa0901889. PMID 19812399
- [Background] van Rees JB, Borleffs CJ, de Bie MK, Stijnen T, van Erven L, Bax JJ, Schalij MJ. Inappropriate implantable cardioverter-defibrillator shocks: incidence, predictors, and impact on mortality. J Am Coll Cardiol. 2011 Feb 1;57(5):556-62. doi: 10.1016/j.jacc.2010.06.059. PMID 21272746
- [Background] Poole JE, Johnson GW, Hellkamp AS, Anderson J, Callans DJ, Raitt MH, Reddy RK, Marchlinski FE, Yee R, Guarnieri T, Talajic M, Wilber DJ, Fishbein DP, Packer DL, Mark DB, Lee KL, Bardy GH. Prognostic importance of defibrillator shocks in patients with heart failure. N Engl J Med. 2008 Sep 4;359(10):1009-17. doi: 10.1056/NEJMoa071098. PMID 18768944
- [Background] Abello M, Merino JL, Peinado R, Gnoatto M, Arias MA, Gonzalez-Vasserot M, Sobrino JA. Syncope following cardioverter defibrillator implantation in patients with spontaneous syncopal monomorphic ventricular tachycardia. Eur Heart J. 2006 Jan;27(1):89-95. doi: 10.1093/eurheartj/ehi500. Epub 2005 Sep 23. PMID 16183691
- [Background] Goldenberg I, Vyas AK, Hall WJ, Moss AJ, Wang H, He H, Zareba W, McNitt S, Andrews ML; MADIT-II Investigators. Risk stratification for primary implantation of a cardioverter-defibrillator in patients with ischemic left ventricular dysfunction. J Am Coll Cardiol. 2008 Jan 22;51(3):288-96. doi: 10.1016/j.jacc.2007.08.058. PMID 18206738
- [Background] Barsheshet A, Moss AJ, Huang DT, McNitt S, Zareba W, Goldenberg I. Applicability of a risk score for prediction of the long-term (8-year) benefit of the implantable cardioverter-defibrillator. J Am Coll Cardiol. 2012 Jun 5;59(23):2075-9. doi: 10.1016/j.jacc.2012.02.036. PMID 22651863
- [Background] Tung R, Josephson ME, Reddy V, Reynolds MR; SMASH-VT Investigators. Influence of clinical and procedural predictors on ventricular tachycardia ablation outcomes: an analysis from the substrate mapping and ablation in Sinus Rhythm to Halt Ventricular Tachycardia Trial (SMASH-VT). J Cardiovasc Electrophysiol. 2010 Jul;21(7):799-803. doi: 10.1111/j.1540-8167.2009.01705.x. Epub 2010 Feb 1. PMID 20132389
- [Background] Hayashi T, Fukamizu S, Hojo R, Komiyama K, Tanabe Y, Tejima T, Soejima K, Nishizaki M, Hiraoka M, Ako J, Momomura S, Sakurada H. Prophylactic catheter ablation for induced monomorphic ventricular tachycardia in patients with implantable cardioverter defibrillators as primary prevention. Europace. 2013 Oct;15(10):1507-15. doi: 10.1093/europace/eut050. Epub 2013 Apr 19. PMID 23603305
- [Background] Dagres N, Cantu F, Geelen P, Lewalter T, Proclemer A, Blomstrom-Lundqvist C. Current practice of ventricular tachycardia ablation in patients with implantable cardioverter-defibrillators. Europace. 2012 Jan;14(1):135-7. doi: 10.1093/europace/eur411. PMID 22167388
- [Background] Horowitz LN, Josephson ME, Farshidi A, Spielman SR, Michelson EL, Greenspan AM. Recurrent sustained ventricular tachycardia 3. Role of the electrophysiologic study in selection of antiarrhythmic regimens. Circulation. 1978 Dec;58(6):986-97. doi: 10.1161/01.cir.58.6.986. PMID 709782
- [Background] Behr ER, Elliott P, McKenna WJ. Role of invasive EP testing in the evaluation and management of hypertrophic cardiomyopathy. Card Electrophysiol Rev. 2002 Dec;6(4):482-6. doi: 10.1023/a:1021161114347. PMID 12438832
- [Background] Kleiman RB, Callans DJ, Hook BG, Marchlinski FE. Effectiveness of noninvasive programmed stimulation for initiating ventricular tachyarrhythmias in patients with third-generation implantable cardioverter defibrillators. Pacing Clin Electrophysiol. 1994 Sep;17(9):1462-8. doi: 10.1111/j.1540-8159.1994.tb01510.x. PMID 7991416
- [Background] Frankel DS, Mountantonakis SE, Zado ES, Anter E, Bala R, Cooper JM, Deo R, Dixit S, Epstein AE, Garcia FC, Gerstenfeld EP, Hutchinson MD, Lin D, Patel VV, Riley MP, Robinson MR, Tzou WS, Verdino RJ, Callans DJ, Marchlinski FE. Noninvasive programmed ventricular stimulation early after ventricular tachycardia ablation to predict risk of late recurrence. J Am Coll Cardiol. 2012 Apr 24;59(17):1529-35. doi: 10.1016/j.jacc.2012.01.026. PMID 22516442
- [Background] Bhavnani SP, Kluger J, Coleman CI, White CM, Guertin D, Shafi NA, Yarlagadda RK, Clyne CA. The prognostic impact of shocks for clinical and induced arrhythmias on morbidity and mortality among patients with implantable cardioverter-defibrillators. Heart Rhythm. 2010 Jun;7(6):755-60. doi: 10.1016/j.hrthm.2010.02.039. Epub 2010 Mar 6. PMID 20211275
- [Background] Costeas XF, Link MS, Foote CB, Homoud MK, Wang PJ, Estes NA. Predictors of ventricular tachycardia recurrence in 100 patients receiving tiered therapy defibrillators. Clin Cardiol. 2000 Nov;23(11):852-6. doi: 10.1002/clc.4960231113. PMID 11097134
- [Background] Daubert JP, Winters SL, Subacius H, Berger RD, Ellenbogen KA, Taylor SG, Schaechter A, Howard A, Kadish A; Defibrillators In Nonischemic Cardiomyopathy Treatment Evaluation (DEFINITE) Investigators. Ventricular arrhythmia inducibility predicts subsequent ICD activation in nonischemic cardiomyopathy patients: a DEFINITE substudy. Pacing Clin Electrophysiol. 2009 Jun;32(6):755-61. doi: 10.1111/j.1540-8159.2009.02362.x. PMID 19545338
- [Background] Zehender M, Brugada P, Geibel A, Waldecker B, Stevenson W, Wellens HJ. Programmed electrical stimulation in healed myocardial infarction using a standardized ventricular stimulation protocol. Am J Cardiol. 1987 Mar 1;59(6):578-85. doi: 10.1016/0002-9149(87)91173-8. PMID 3825897
- [Background] Kulakowski P, Bashir Y, Heald S, Paul V, Anderson MH, Gibson S, Malik M, Camm AJ. Effects of procainamide on the signal-averaged electrocardiogram in relation to the results of programmed ventricular stimulation in patients with sustained monomorphic ventricular tachycardia. J Am Coll Cardiol. 1993 May;21(6):1428-39. doi: 10.1016/0735-1097(93)90320-z. PMID 8473652
- [Background] Kuller L, Lilienfeld A, Fisher R. An epidemiological study of sudden and unexpected deaths in adults. Medicine (Baltimore). 1967 Jul;46(4):341-61. doi: 10.1097/00005792-196707000-00003. No abstract available. PMID 6043997
- [Derived] Futyma P, Futyma M, Kulakowski P. Non-invasive programmed stimulation to identify high-risk patients with implanted cardioverter defibrillator (the NIPS-ICD study): study protocol for a randomized controlled trial. Trials. 2016 Jan 27;17:50. doi: 10.1186/s13063-016-1170-2. PMID 26818636